CLINICAL TRIAL: NCT05510687
Title: A Randomised Controlled Trial on the Impact of Free Reading Glasses to Support Use of Smartphone Banking in Bangladesh Among Government Old Age Allowance and Widow Allowance Beneficiaries
Brief Title: Transforming Households With Refraction and Innovative Financial Technology
Acronym: THRIFT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: L.V. Prasad Eye Institute (Other); VisionSpring (Other); MOMODa Foundation (Unknown); Good Business Labs Foundation (Unknown); Florida International University (Other); Clearly (Other); BRAC University (Other)
Responsible Party: Principal Investigator, Nathan Congdon, Principal Investigator, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MHLS 22_69
Record Dates: First submitted 2022-08-18; First posted 2022-08-22 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Presbyopia
Keywords: Presbyopia; Digital transactions and vision
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Intervention Model Description: THRIFT is a randomised controlled trial (RCT) that employs an explanatory embedded mixed methods design whereby the RCT is the primary study, and the secondary or embedded approach is a mixed-methods investigation of the culture and context surrounding the trial. The basic RCT design employs individual OAA and WA beneficiary-households in digitised safety-net catchment areas as the unit of randomization. The study uses a two-arm RCT design, one treatment and one control arm. Only households with an eligible participant who does not personally own a smartphone or feature phone and .access DFS through any phone during the time of the trial. The duration of the RCT is 18 months. The trial will be investigator masked.
Who Masked: Investigator
Masking Description: The trial will be investigator-masked, but Community Health Workers (CHW), other fieldwork personnel and the participants will not be masked to Intervention Group assignment. This is because participants in the Intervention Group will receive eyeglasses at the start of the trial and members of the Control Group will receive theirs at the end. All care will be taken to ensure that the investigators who are not involved in fieldwork will be kept masked, and they do not foresee conditions that will require emergency unmasking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glasses to correct presbyopia and digital financial training (Experimental): The intervention is the provision of glasses to correct presbyopia plus digital financial training to use bKash, a popular mobile banking application that is becoming the preferred mode of transferring payments to the bank accounts of OAA and WA beneficiaries in Bangladesh.
  Interventions: Device: Glasses to correct presbyopia
- Control-No treatment (No Intervention): Mobile phone with preloaded bank transaction tracking app: Participants will be provided a basic mobile phone handset. The bank transaction tracking application that is being developed to measure the primary outcomes for this trial will be installed on these phones before giving them to the participants. A mobile data pack will also be remotely loaded on the mobile phone to facilitate internet access for mobile banking.
  Eyeglasses: These participants will receive a free pair of eyeglasses at the conclusion of the study to correct refractive errors, unless they have obtained such glasses on their own during the study.

INTERVENTIONS:
Device: Glasses to correct presbyopia — Participants will receive eyeglasses to correct presbyopia, as per the power determined in the eye examination.
  Arms: Glasses to correct presbyopia and digital financial training

SUMMARY:
The aim of the proposed Randomised Clinical Trial (RCT) is to assess the impact of presbyopia correction and basic digital financial training on greater adoption and use of digital financial services (primary outcome) and other welfare impacts (secondary outcomes)) for safety-net beneficiaries in Bangladesh. Trial participants will be Old Age Allowance (OAA) and Widows Allowance (WA) beneficiaries who regularly receive payments as part of a government safety net program for the very poor.

The primary objective of the THRIFT trial is to assess whether the combined complementary intervention of providing free eyeglasses and basic digital financial services training in the use of mobile phones to recipients of government OAA and WA safety-net payments can lead to greater financial inclusion and improved quality of life.

THRIFT's primary outcome is the adoption and effective use of the DFS platform in receiving digital OAA and WA transfers using the mobile banking platform, as measured by the difference between the treatment and control groups.

The secondary outcomes analysed under the THRIFT trial will be:

total data consumption, independent use of the mobile banking application, purchase of eyeglasses (for control group members), access to medication and healthcare, subjective well-being, mobility, social connectedness, percentage of household consumption, reasons for using or avoiding smartphone based DFS, and decision-making power within the household.

DETAILED DESCRIPTION:
Background and Rationale: The proliferation of mobile banking systems across developing countries has provided previously un-banked populations with a convenient method to manage their finances digitally. The Government of Bangladesh launched the Old Age Allowance (OAA) and Widow Allowance (WA) programmes in 1998 to provide a financial safety net to its poor and vulnerable population - elderly under OAA and vulnerable women under WA. More than half of Bangladesh adults lack access to a formal bank account, with most of the un-banked population belonging to the poorest 40% of households. Mobile money, through applications such as bKash, has become the "innovation" to improve the financial inclusion scenario in Bangladesh, especially during the coronavirus pandemic. The take-up of mobile money is often limited by a lack of technical awareness and trust concerns among the elderly. Lee at al. (2021) have addressed these concerns through an intervention consisting of initial training and subsequent minor assistance in using the bKash mobile banking application, which they randomised over a sample of poor households in rural Bangladesh. They found an increase of 7.5% in rural consumption, a reduction in extreme poverty and a 26% increase in urban to rural remittances among the sample participants using bKash a year after the intervention. Across Low and Middle Income Countries (LMICs), experimental studies encouraging adoption of mobile money applications have been shown to improve consumption smoothing, savings and access to credit. There is evidence to support the theory that a training module introducing the elderly to mobile banking will help bridge strong information and trust gaps, and encourage greater financial independence. As traditional joint family structures weaken in South Asian societies, greater economic independence among older populations has the potential to improve their functional independence, level of healthcare access, and mental well-being. Evidence suggests that there is a substantial burden of uncorrected presbyopia in Bangladesh. Uncorrected vision problems have been found to negatively affect visual function, which includes smart phone and mobile phone usage among the elderly in multiple LMIC contexts. It has also been found to affect productivity among tea plantation workers performing visually demanding tasks in Assam, India. This can lead to lower engagement with mobile banking platforms, which in turn can limit elderly people's access to their finances. Conversely, correction of presbyopia is associated with significant improvements in work productivity and other economically important outcomes.

The proposed THRIFT trial is the first randomised trial to examine two important determinants of mobile banking among an elderly and financially vulnerable population in a developing country context: lack of awareness about the use of mobile banking, and uncorrected age-related decline in near vision, presbyopia.

The aim of the proposed RCT trial is to assess the impact of presbyopia correction and basic digital financial training (combined complementary intervention) on greater adoption and use of digital financial services (primary outcome) and other welfare impacts (secondary outcomes) for safety-net beneficiaries in an LMIC.

JPGSPH will gather the beneficiary list of the OAA and WA from the Department of Social Service, Government of Bangladesh.

Consent for Social screening and vision screening is obtained by Community Health workers (CHW) of MOMODa Foundation (MF) and consented participants are assigned the Unique participant Identifier (ID).

All the relevant documents are verified before proceeding to the social screening.

Social screening including numeracy, dexterity and cognitive test (NDC test) is done to confirm eligibility.

Eligible participant list is shared with VisionSpring (VS) team after obtaining consent for vision examinations.

VS CHWs and Programs officers conduct door-to door eye-screening for presbyopia diagnosis and eligible participant list is shared with MF for proceeding with baseline survey. Consent for baseline survey and trial is obtained by MF, followed by randomisation.

Treatment group gets the eyeglasses, mobile phone and basic training on the usage of the mobile phone and mobile banking application.

Control group gets mobile phone and basic instructions to use the mobile phone and prescription for glasses. Eyeglasses to the control group are provided at the end of the study.

VS team conducts 2 follow up visits per participant, one month and 6 months after receiving glasses with a one month additional window for each visit.

* to check the compliance to eyeglasses
* Collect any safety event information MOMODa Foundation team conducts 2 follow-up visits per participant at 3 and 6 months after providing the smartphones and training with a one month additional window for each visit.If it is not possible to meet during that window period, the survey will be completed by telephonic survey within the next 7 days after the allowed one-month window. MF
* collects any information on safety events
* checks the smartphones provided
* assesses the participants comfort to use the smartphone
* assesses whether smartphone is being used by the participant. MF conducts the endline survey 18 months after the distribution of the smartphones.

Study Setting:

The research will be conducted in Kurigram Sadar and Nageshwari, two sub-districts within the Kurigram district located in northern Bangladesh. These districts are in bKash catchment area for the Department of Social Services safety-net payments. Specifically, the study will take place in nine unions, seven in Kurigram Sadar and two in Nageshwari.

Recruitment: This will begin with the receipt of the list identifying OAA and WA beneficiaries living in Kurigram district from the Department of Social Service, Government of Bangladesh.

Before visiting the beneficiaries' households, the enumerators will make phone calls to schedule appointments.

MF will conduct a door-to-door social screening survey based on the eligibility criteria.

Numeracy, Dexterity and Cognition (NDC) Test: The study participants who will meet all inclusion criteria up to this point and attended the Social Screening Survey will undergo a basic numeracy and a functional literacy test. This is to assess if they can conduct basic operations using a phone, such as recognising numbers and using the smartphone screen number pad to enter numbers.

Before conducting the social screening survey and NDC test, beneficiaries will be requested to familiarise themselves with the numbers (English) from 0 to 9 prior to the scheduled household visit.

During this test, beneficiaries will be requested if they can see the numbers on app and based on the visual demand they will be given +1, +2 or +3 reading glasses starting with +1 for 48-50 age group, +2 for 51-60 age group, and +3 >60 age.

Presbyopia diagnosis: Door-to-door eye screening examinations will be done to all the identified OAA and WA beneficiaries in the selected district who consent to be screened.

Baseline Survey: After undergoing social screening, NDC test, and vision screening, the individuals will be selected for the baseline survey.

RANDOMISATION AND PROCEDURES Participants will be randomly assigned to either the Intervention or Control Group using following procedure.

The randomization sequence will be generated by the study statistician at the L.V. Prasad Eye Institute Clinical Trials Unit (LVPEI CTU) using a pre-written code in Stata. Separate randomisation sequences will be prepared in advance for each of the 12 possible strata.

Allocation concealment mechanism The allocation sequence will be in a password protected location stored in designated folder for THRIFT by James P Grant School of public Health (JPGSPH) and will be accessed by the concealment implementers only.

The implementation team will receive a list of beneficiaries and their respective group allocation based on the baseline data collected. The group allocation for a participant will be revealed from the list and the participant is enrolled.

Blinding/Masking The trial will be investigator-masked, but CHWs, other fieldwork personnel and the participants will not be masked to Intervention Group assignment.

ANALYSIS Baseline demographic and clinical characteristics will be reported for all participants in the sample, excluding protocol deviations randomised in error where Informed Consent has not been obtained. Baseline characteristics will be summarised by their means and standard deviations, medians and interquartile ranges, or numbers and percentages as appropriate.

An intention to treat (ITT) approach will be used to analyse the trial outcomes. This will involve regressing the outcome of concern on the randomised intervention status, difference in differences (DID) for panel data will be used for analysis. The primary analysis will be stratified by (1) WA recipients vs OAA recipients (2) incoming vs. outgoing transactions, and (3) smartphone-based vs. non-smartphone-based transactions (e.. kiosk use). All analyses will be adjusted for age, gender, and previous phone use. Random imbalances may occur hence, both the crude and adjusted estimates will be presented, but the primary inference will be based on the adjusted analysis. Several studies with regional and rural samples have found vision problems to affect ageing populations in Bangladesh. Previously, there has been a gender gap in eye health in Bangladesh. In 2023, Orbis, the Fred Hollows Foundation and its partners started work to close this gap. Uncorrected vision problems have been found to negatively affect visual function, for example, smartphone and mobile phone usage among the elderly in multiple LMIC contexts.The rates of mobile banking usage, as measured in the primary outcomes, will be compared across groups of participants based on the basis of age, education, household income and other socioeconomic variables. Standard errors will be clustered at the individual level for this analysis. However, for high-frequency outcome variables (such as app-based financial transactions) data will be aggregated at the appropriate level (either monthly or weekly or quarterly), with errors clustered at the household level. Outcome variables that are binary in nature will be analysed using Linear Probability Model Method.

Participants will be described with respect to the following characteristics at trial entry:

Age, Sex, Education level, Uncorrected, presenting and corrected distance visual acuity in each eye separately and both eyes together, Ownership of glasses for the correction of distance vision and self-reported regularity of use Visual Function Questionnaire (VFQ-25), Rural residence, Attitudes towards vision correction, Access to local eye care services, history of uptake of eye care services.

Numbers (with percentages) for binary and categorical variables and means (and standard deviations), or medians (with lower and upper quartiles) for continuous variables will be presented; there will be no tests of statistical significance performed nor confidence intervals calculated for differences between groups on any baseline variables (for instance mid-way through trial from Interim Analysis).

Economic Evaluation An economic evaluation of the intervention will be conducted using cost-effectiveness analysis. Data will be collected on the incremental cost of providing eyeglasses to the Intervention Group to calculate the incremental cost per quality-of-life measure, which will help assess the cost-effectiveness of the intervention.

No planned interim analysis will be undertaken due to the short duration of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age

   * 65-70 years old male OAA beneficiaries
   * 62-70 years old female OAA beneficiaries
   * 48-60 years old WA beneficiaries
2. Receiving digital OAA or WA payments from the Government of Bangladesh
3. Residence Lived in the bKash catchment area, Kurigram for 3 more
4. Presbyopia

   * Binocular presenting near-vision N6.3 or worse, correctable to N5 or better
   * Require a new pair of glasses
5. Mapped into bottom three asset quintiles according to the equity tool questionnaire
6. Numeracy, dexterity and cognitive ability Score 8 or above on NDC Screening test.
7. Individuals who do not use Mobile Financial Services (MFS) account by themselves

Exclusion criteria

1. Poor internet connection, less than 13kbps
2. Presence of any cause of near or distance vision impairment that cannot be resolved with presbyopic glasses.

Ages: 48 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 571 (Actual)
Dates: Start 2023-12-10 (Actual); Primary Completion 2025-09-08 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change in the average number, difference in the mean value, difference in the mean total value of transactions per participant per quarter comparing a 12-month period before the intervention to a 18-month period after the intervention | Once every quarter through study completion (up to 18 months)
  This will be calculated using both the incoming and outgoing transaction level data from bKash.

SECONDARY OUTCOMES:
Application was facilitated by a bKash agent or family member, or independently by the beneficiary. | Change from baseline to 18 months
  Whether use of the application was facilitated by a bKash agent or family member, or independently by the beneficiary. This will be collected using the baseline and endline surveys developed for the trial. Categorical
Purchase of additional phones by study participant's household | Change from baseline to 18 months
  Purchase of additional phones per household is assessed using the endline survey. Any purchase recorded with either Yes or No
Purchase of additional phones by study participant | Change from baseline to 18 months
  Purchase of additional phones by the individual is assessed using the endline survey. Any purchase recorded with either Yes or No
Intra-household resource sharing by the beneficiary | Change from baseline to 18 months
  Percentage of resource shared by the beneficiary from total household consumption is assessed using the survey instrument developed for the trial. Best score is 100 and worst score is 0.
Purchase of glasses other than those issued to the intervention group | Change from baseline to 18 months
  Glasses purchased by the study participant is assessed using the endline survey instrument developed for the trial. A binary outcome with either Yes or No.
Food security | Up to 18 months
  Participants perception of the nutrition and quantity of their daily food consumption is measured using standard module developed by World Food Programme (WFP). This is a categorical (mild, moderate, severe) index with larger values indicating higher levels of food insecurity.
Role of study participant in household decision making autonomy | Change from baseline to 18 months
  The onus of decision making for different household activities by the participant is assessed using the baseline and endline survey instruments developed fort the trial. Best score is 100% and worst score is 0%
Subjective well-being of study participants, quality of life | Change from baseline to 18 months
  Participants satisfaction with various aspects of their life such as personal relationships is assessed using the Quality of Life survey EuroQoL-5 Dimesions-5Levels(EQ-5D-5L). Best score is 100 and worst score is 0.
Subjective well-being of study participants, vision assessment | Change from baseline to 18 months
  Participants satisfaction with various aspects of their life such as their health is assessed using the Near Activity Visual Questionnaire (NAVQ). Best score is 100 and worst score is 0.
Mobility of study participant | change from baseline to18 months
  Participants comfort in regular physical activities is assessed using International Physical Activity questionnaire (IPAQ) is collected at baseline and endline.
Social connectedness of study participant | Change from baseline to 18 months
  Participants engagement with their family members, friends and neighbors is assessed using baseline and endline surveys. The best possible score is 12 and the worst possible score is 0.
Reasons for uptake or avoidance of smartphone based DFS. | Once every quarter through study completion (up to 18 months)
  Reasons for using or avoiding smartphone based DFS among the participants is surveyed and analysed as a categorical outcome.
Incidence of theft or fraudulent use of money | Up to 18 months
  Self-reported incidents on theft from the index participant's bank account using the baseline survey. A binary outcome with either Yes or No
Assessment of depressive disorders | 18 months
  Participants'mental health is assessed using Patient Health Questionnaire 9 during the endline survey as a contiuous variable.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan G Congdon, MD, MPH, Principal Investigator — Queen's University, Belfast; Atonu Rabbani, PhD, Principal Investigator — BRAC James P Grant School of Public Health; Abu S Shonchoy, PhD, Principal Investigator — Florida International University
Locations (1):
- James P. Grant School of Public Health BRAC University, Dhaka, Bir Uttom A K Khandakar Road, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
All Individual Participant Data (IPD) will be stored in anonymised format. The IPD that includes personal identifiable information will be deleted when the data collection process is complete and before the initiation of data analysis.
  Only de-identified data will be shared with all the researchers for analysis. The primary analysis will be conducted on all outcome data obtained from all enrolled participants as randomised.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: All deidentified IPD will be available from January 2023 (anticipated Trial start date) to Aug 2024 (inclusive of analysis, report writing and publication).
Access Criteria: Following publication of the primary and secondary outcomes there may be scope to conduct additional analyses on the data collected. In such instances formal requests for data will need to be made in writing to the Chief Investigator, who will discuss this with the Sponsor. The study will comply with the good practice principles for sharing individual participant data from publicly funded clinical trials and data sharing will be undertaken in accordance with the required regulatory requirements.

REFERENCES:
- [Background] Suri T, Jack W. The long-run poverty and gender impacts of mobile money. Science. 2016 Dec 9;354(6317):1288-1292. doi: 10.1126/science.aah5309. Epub 2016 Dec 8. PMID 27940873
- [Background] Khanam MA, Streatfield PK, Kabir ZN, Qiu C, Cornelius C, Wahlin A. Prevalence and patterns of multimorbidity among elderly people in rural Bangladesh: a cross-sectional study. J Health Popul Nutr. 2011 Aug;29(4):406-14. doi: 10.3329/jhpn.v29i4.8458. PMID 21957680
- [Background] Lu Q, Congdon N, He X, Murthy GV, Yang A, He W. Quality of life and near vision impairment due to functional presbyopia among rural Chinese adults. Invest Ophthalmol Vis Sci. 2011 Jun 13;52(7):4118-23. doi: 10.1167/iovs.10-6353. PMID 21508106
- [Background] Patel I, Munoz B, Burke AG, Kayongoya A, McHiwa W, Schwarzwalder AW, West SK. Impact of presbyopia on quality of life in a rural African setting. Ophthalmology. 2006 May;113(5):728-34. doi: 10.1016/j.ophtha.2006.01.028. PMID 16650665
- [Background] Rahman FN, Khan HTA, Hossain MJ, Iwuagwu AO. Health and wellbeing of indigenous older adults living in the tea gardens of Bangladesh. PLoS One. 2021 Mar 4;16(3):e0247957. doi: 10.1371/journal.pone.0247957. eCollection 2021. PMID 33662034
- [Background] Laviers H. The prevalence of presbyopia and the feasibility of community distribution of near spectacles in adults in Zanzibar, East Africa. Community Eye Health. 2007 Dec;20(64):73. No abstract available. PMID 18330449
- [Background] Wang C, Wang X, Jin L, Tang B, Zhu W, Zhang G, Chen T, McAneney H, Kassalow J, Congdon N. Influence of presbyopia on smartphone usage among Chinese adults: A population study. Clin Exp Ophthalmol. 2019 Sep;47(7):909-917. doi: 10.1111/ceo.13559. Epub 2019 Jun 13. PMID 31090978
- [Background] Mathieson KM, Kronenfeld JJ, Keith VM. Maintaining functional independence in elderly adults: the roles of health status and financial resources in predicting home modifications and use of mobility equipment. Gerontologist. 2002 Feb;42(1):24-31. doi: 10.1093/geront/42.1.24. PMID 11815696
- [Background] Srivastava S, Purkayastha N, Chaurasia H, Muhammad T. Socioeconomic inequality in psychological distress among older adults in India: a decomposition analysis. BMC Psychiatry. 2021 Apr 7;21(1):179. doi: 10.1186/s12888-021-03192-4. PMID 33823847
- [Background] Muhit M, Minto H, Parvin A, Jadoon MZ, Islam J, Yasmin S, Khandaker G. Prevalence of refractive error, presbyopia, and unmet need of spectacle coverage in a northern district of Bangladesh: Rapid Assessment of Refractive Error study. Ophthalmic Epidemiol. 2018 Apr;25(2):126-132. doi: 10.1080/09286586.2017.1370119. Epub 2017 Oct 4. PMID 28976783
- [Background] Muhammad N, Alhassan MB, Umar MM. Visual function and vision-related quality of life in presbyopic adult population of Northwestern Nigeria. Niger Med J. 2015 Sep-Oct;56(5):317-22. doi: 10.4103/0300-1652.170379. PMID 26778881
- [Background] Jack, W., & Suri, T. (2014). Risk Sharing and Transactions Costs: Evidence from Kenya's Mobile Money Revolution. American Economic Review, 104(1), 183-223. https://doi.org/10.1257/aer.104.1.183
- [Background] Kidd Man RE, Fenwick EK, Sabanayagam C, Li LJ, Gupta P, Tham YC, Wong TY, Cheng CY, Lamoureux EL. Prevalence, Correlates, and Impact of Uncorrected Presbyopia in a Multiethnic Asian Population. Am J Ophthalmol. 2016 Aug;168:191-200. doi: 10.1016/j.ajo.2016.05.019. Epub 2016 May 28. PMID 27246256
- [Background] Reddy PA, Congdon N, MacKenzie G, Gogate P, Wen Q, Jan C, Clarke M, Kassalow J, Gudwin E, O'Neill C, Jin L, Tang J, Bassett K, Cherwek DH, Ali R. Effect of providing near glasses on productivity among rural Indian tea workers with presbyopia (PROSPER): a randomised trial. Lancet Glob Health. 2018 Sep;6(9):e1019-e1027. doi: 10.1016/S2214-109X(18)30329-2. Epub 2018 Jul 23. PMID 30049615
- [Background] Aker, J., & Mbiti, I. (2010). Mobile Phones and Economic Development in Africa. Journal Of Economic Perspectives, 24(3), 207-232. https://doi.org/10.1257/jep.24.3.207
- [Background] Bangladesh Bureau Of Statistics, Statistics and Informatic Division, Ministry of Planning. Government of Bangladesh. (2015). Age-Sex Composition of Bangladesh Population. http://203.112.218.65:8008/WebTestApplication/userfiles/Image/PopMonographs/Volume-9_Age-Sex.pdf
- [Background] Chiroma, M., & Jamda, A. (2017). Impact of Uncorrected Presbyopia on the Quality of Life in Rural Gwagwalada, Nigeria. Journal Of Community Medicine And Primary Health Care, 29(1). 15 October 2021 https://www.ajol.info/index.php/jcmphc/article/view/160834
- [Background] Kabir, R., T.A.Khan, H., Kabir, M., & Rahman, M. (2013). POPULATION AGEING IN BANGLADESH AND ITS IMPLICATION ON HEALTH CARE. European Scientific Journal, 9(33). Retrieved 15 October 2021, from https://core.ac.uk/download/pdf/83951388.pdf
- [Background] Khan, M., Islam Mondal, M., Hoque, N., & Islam, M. (2014). A Study on Quality of Life of Elderly Population in Bangladesh. American Journal Of Health Research, 2(4), 152. https://doi.org/10.11648/j.ajhr.20140204.18
- [Background] World Bank. (2018). Br Project Appraisal Document On A Proposed Credit In The Amount Of Sdr 213.60 Million (Us$ 300.00 Million Equivalent) To The People's Republic Of Bangladesh For A Cash Transfer Modernization Project. World Bank. Retrieved from https://documents1.worldbank.org/curated/en/258451517626830719/pdf/BANGLADESH-PAD-01112018.pdf
- [Background] Baur-Yazbeck, S. (2019). A New Generation of Government-to-Person Payments Is Emerging. CGAP. Retrieved 15 October 2021 https://www.cgap.org/blog/new-generation-government-person-payments-emerging
- [Background] Shonchoy, A., Rigol, N., Roth, B., Chandra, S., Franco, A., & Hussam, R. (2021). Safety Nets and the Pandemic: The State of Social Benefit Payments during COVID-19. Unpublished manuscript https://poverty-action.org/sites/default/files/The%20State%20of%20Social%20Benefit%20Payments%20in%20Bangladesh%20during%20COVID-19.pdf
- [Background] World Bank Group. "PROGRAM BRIEF: Old Age Allowance." worldbank.org, 2019 https://documents1.worldbank.org/curated/en/619861552541446911/pdf/135280-13-3-2019-9-14-4-ProgrambriefonOAAF.pdf
- [Background] World Bank. (2017). Chapter 2: The Unbanked. https://globalfindex.worldbank.org/sites/globalfindex/files/chapters/2017%20Findex%20full%20report_chapter2.pdf
- [Background] Khatun, M., Mitra, S., & Sarkar, M. (2021). Mobile banking during COVID-19 pandemic in Bangladesh: A novel mechanism to change and accelerate people's financial access. Green Finance, Aims Press, 3(3), 253-267. Retrieved 15 October 2021, from https://www.aimspress.com/article/doi/10.3934/GF.2021013?viewType=HTML
- [Background] Msweli, N., & Mawela, T. (2020). Enablers and Barriers for Mobile Commerce and Banking Services Among the Elderly in Developing Countries: A Systematic Review. Lecture Notes In Computer Science, 319-330. https://doi.org/10.1007/978-3-030-45002-1_27
- [Background] Rajaobelina, L., Brun, I., Line, R. and Cloutier-Bilodeau, C. (2021), Not all elderly are the same: fostering trust through mobile banking service experience, International Journal of Bank Marketing, Vol. 39 No. 1, pp. 85-106. https://doi.org/10.1108/IJBM-05-2020-0288
- [Background] Lee, J., Morduch, J., Ravindran, S., Shonchoy, A., & Zaman, H. (2021). Poverty and Migration in the Digital Age: Experimental Evidence on Mobile Banking in Bangladesh. American Economic Journal: Applied Economics, 13(1), 38-71. https://doi.org/10.1257/app.20190067
- [Background] Aker, J., Boumnijel, R., McClelland, A., & Tierney, N. (2016). Payment Mechanisms and Antipoverty Programs: Evidence from a Mobile Money Cash Transfer Experiment in Niger. Economic Development And Cultural Change, 65(1), 1-37. https://doi.org/10.1086/687578
- [Background] Catia Batista & Pedro C. Vicente, 2018.
- [Background] Bastian, G., Bianchi, I., Goldstein, M., & Montalvao, J. (2021). Short-Term Impacts of Improved Access to Mobile Savings, with and without Business Training: Experimental Evidence from Tanzania - Working Paper 478. Center For Global Development. Retrieved 15 October 2021 https://www.cgdev.org/publication/short-term-impacts-improved-access-mobile-savings-business-training
- [Background] Riley, E. (2018). Mobile money and risk sharing against village shocks. Journal Of Development Economics, 135, 43-58. https://doi.org/10.1016/j.jdeveco. 2018.06.015
- [Background] Goli, S., Reddy, B., Srinivasan, V., & James, K. (2019). Economic Independence and Social Security among India's Elderly. Economic And Political Weekly, 39. Retrieved 15 October 2021
- [Background] Hamiduzzaman, M., de Bellis, A., Abigail, W., & Kalaitzidis, E. (2018). Elderly Women in Rural Bangladesh. South Asia Research, 38(2), 113-129. https://doi.org/10.1177/0262728018767018
- [Background] World Bank Group. "PROGRAM BRIEF: Allowances for the Widow, Deserted and Destitute Women" worldbank.org, 2019 https://documents1.worldbank.org/curated/en/994221552537440138/pdf/135277-BRI-PUBLIC-13-3-2019-9-15-58-ProgrambriefonWAF.pdf
- [Background] Basic and Clinical Science Course, Section 03: Clinical Optics and Vision Rehabilitation. (n.d.). https://store.aao.org/basic-and-clinical-science-course-section-03-clinical-optics-and-vision-rehabilitation.html
- [Background] Bangladesh Bureau of Statistics. Household Income & Expenditure Survey 2016. Dhaka; 2017.
- [Background] Food Insecurity Experience Scale (FIES) |Policy Support and Governance| Food and Agriculture Organization of the United Nations. (n.d.) https://www.fao.org/policy-support/tools-and-publications/resources-details/en/c/1236494/
- [Background] World Food Program. Food Security and Nutrition Assessment. 2019; https://docs.wfp.org/api/documents/WFP-0000108055/download/
- [Background] Devlin N, Pickard S, Busschbach J. The Development of the EQ-5D-5L and its Value Sets. 2022 Mar 24. In: Devlin N, Roudijk B, Ludwig K, editors. Value Sets for EQ-5D-5L: A Compendium, Comparative Review & User Guide [Internet]. Cham (CH): Springer; 2022. Chapter 1. Available from http://www.ncbi.nlm.nih.gov/books/NBK589306/ PMID 36810043
- [Background] Sharma G, Chiva-Razavi S, Viriato D, Naujoks C, Patalano F, Bentley S, Findley A, Johnson C, Arbuckle R, Wolffsohn J. Patient-reported outcome measures in presbyopia: a literature review. BMJ Open Ophthalmol. 2020 Jul 12;5(1):e000453. doi: 10.1136/bmjophth-2020-000453. eCollection 2020. PMID 32685693
- [Background] Gupta N, Wolffsohn JS, Naroo SA, Davies LN, Gibson GA, Shah S. Development of a near activity visual questionnaire to assess accommodating intraocular lenses. Cont Lens Anterior Eye. 2007 May;30(2):134-43. doi: 10.1016/j.clae.2007.01.004. Epub 2007 Feb 26. PMID 17324609
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Cohen S, Doyle WJ, Skoner DP, Rabin BS, Gwaltney JM Jr. Social ties and susceptibility to the common cold. JAMA. 1997 Jun 25;277(24):1940-4. PMID 9200634
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Derived] Shitol SA, Aftab IB, Piyasena P, Lohfeld L, Rayasam S, Challa N, Sangani P, Sigwadhi LN, Rahman HMM, Khanna RC, Chan VF, Barua M, Pant S, Adhvaryu A, Nyshadham A, Sarker M, Mettla AL, Haque E, MacKenzie G, Alam S, Gudwin E, Clarke M, Shonchoy A, Rabbani A, Congdon N. Transforming Households with Refraction and Innovative Financial Technology (THRIFT): study protocol for a randomised controlled trial of vision interventions and online banking among the elderly in Kurigram. BMJ Open. 2024 Dec 23;14(12):e085083. doi: 10.1136/bmjopen-2024-085083. PMID 39719288
- See also: The Fred Hollows Foundation. (2023). Closing the gender gap in eye health in Bangladesh — https://www.hollows.org/en-US/latest-news/closing-the-gender-gap-in-eye-health-in-bangladesh/
- See also: Orbis International. (2023). Closing the gender gap in eye care across Banglades — https://gbr.orbis.org/en/news/2023/international-womens-day-2023

DOCUMENTS (1):
  • Statistical Analysis Plan (2026-01-25): https://cdn.clinicaltrials.gov/large-docs/87/NCT05510687/SAP_002.pdf